CLINICAL TRIAL: NCT07029841
Title: Cohort Study on Treatment Comes of Catheter-based Therapy in Patients With Acute Pulmonary Embolism in Hong Kong - the HONG KONG PECT Registry
Brief Title: Cohort Study on Treatment Comes of Catheter-based Therapy in Patients With Acute Pulmonary Embolism in Hong Kong
Acronym: HK-PECT
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2022.121; 2022.121 (Other: CUHK-NTEC CREC)
Record Dates: First submitted 2025-06-04; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism Acute; Pulmonary Embolism Acute Massive; Pulmonary Embolism Subacute Massive
Keywords: PE, CDT, LBAT, UACDT
MeSH Terms: conditions — Focal cortical dysplasia of Taylor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- catheter-directed thrombolysis (CDT): Patient treated by any mode of catheter-directed thrombolysis, including ultrasound assisted catheter directed thrombolysis (EKOS).
  Interventions: Device: catheter-based therapy
- Aspiration thrombectomy (AT): Patient treated by any mode of aspiration thrombectomy, including large-bore mechanical thrombectomy (LBMT) such as Penumbra, Flowtriever, or Alphavac.
  Interventions: Device: catheter-based therapy

INTERVENTIONS:
Device: catheter-based therapy — catheter-based therapy

SUMMARY:
This retrospective cohort study (Hong Kong PECT Registry) compares treatment outcomes between different percutaneous catheter-based therapies in patients with acute pulmonary embolism (PE). PE is a critical condition with potential for rapid deterioration and mortality before treatment. While availability of catheter-based therapy contributed to the declining mortality rates of PE, selecting the appropriate intervention remains key. There are primarily two modes of therapies available: Catheter-directed thrombolysis and Aspiration thrombectomy (e.g., Penumbra, Flowtriever, AlphaVac) Given limited direct comparisons between these methods, the study will evaluate their efficacy, safety, and clinical outcomes of these treatment strategies in acute PE patients.

DETAILED DESCRIPTION:
Introduction Acute pulmonary embolism is a well known disease to all cardiologists and physicians. Not only because of the disease is not uncommon, not a small portion of patients suffered from acute pulmonary embolism may deteriorate suddenly and rapidly, before the intiation of treatment. Luckily, time trend analyses throughout the world the mortality of pulmonary embolism is on decreasing trend.

Besides traditional systemic thrombolysis and surgical embolectomy, percutaneous catheter directed treatment has been used recently as well, especially those who are poor surgical candidates while not eligible to systemic thrombolytics. There are different types of percutaneous catheter directed treatment. Boardly can be divided as the catheter interventions with or without use of thrombolysis and catheter based aspiration thrombectomy. In our local experiences, EKOS is one of the example as catheter interventions with the use of thrombolysis, by using ultrasound assisstance. While IndigoVR Mechanical Thrombectomy System (Penumbra), Flowtriever system (Inari) and AlphaVac (angiodynamic) are some of examples of the aspiration thrombectomy.

Direct comparions between different types of percutaneous cathter directed treatment is limited. With the local datas avaliable, we would like to compare the efficacy, safety and other significant clinical outcomes between different types of catheter-based therapies.

Objectives In patient with pulmonary embolism who underwent percutaneous catheter directed treatment , is there any difference interms of clinical efficacy, safety outcomes and other significant clinlcal parameters? Patients and Methods Inclusion criteria

1. Adults >= 18 years
2. Patients who were admitted to Pok Oi Hospital, Tuen Mun Hospital, Prince of Wales Hopstial from Jan 2016 to December 2021 and diagnosed to have acute pulmonary embolism
3. Receiveed treatment of any types of catheter-based therapy for pulmonary embolism Exclusion Criteria

1) no exclusion criteria

As this is an all comers registry, there is no upper limit of sample size. Consent As this retrospective study only involve data collection and no active intervention to the patients, consent will be waivered. Only necessary and relevant existing clinical data will be retirieved by desiganted investigators from electronic medical records stored in the clinical management system of the participating hospitals. Only if necessary (e.g. if data not avaliable in electronic system from clinical management system ) , the kardex will be retrieved and returned as soon as possible Any identifying information will be removed before further storage, and analysis. Data entry, storage, analysis and presentations will be processed anonymously. Confidentiality and ethical use of the data is safeguard with all data only accessible to designated investigators. All the data will be deleted, removed and destroyed after 5 years of study completion.

Potential risk and benefit The major risk to study participants is confidentiality regarding identifiable, private health information - specifically, medical record numbers. To maintain security of this information, the database of included participants will be kept in a password-protected computer with antivirus software within the hospital compound.

Methodology The patients will be searched in hospital authority CMS record with key words Diagnosis Code Acute pulmonary embolism and infarction and procedural code of infusion of thrombolytic agent and incision of other thoracic vessels.

Afterwards the recruited cases will be reviewed , either selected or abandoned according to inclusion and exclusion criteria. This study will be conducted in compliance to the Declaration of Helsinki.

Outcomes Measures With the appropriate cases selected according to inclusion and exclusion criteria, clinical parameters will be reviewed analyzed. in-patient hospitality will be reviewed as primary outcomes. Secondary endpoints include 90 days mortality, 90 days PE related mortality, 90 days PE recurrence, and procedural efficacy outcomes including the change in the right ventricle to left ventricle ratio and mean pulmonary artery pressure. Other safety outcomes or clinical parameters will be also evaluated which include procedural complications, major bleeding events, procedural time, hemoglobin change after procedure, need of blood transfusion and usage of Intravenous fluid in first 72 hours after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is admitted with a diagnosis of acute pulmonary embolism
* Patient who receives any types of catheter-based therapy for acute pulmonary embolism.

Exclusion Criteria:

* nil. This is a all-comer registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry aims to evaluate the efficacy and safety of patients with acute PE treated with catheter-based therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2032-12-28 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Inpatient mortality rates | baseline, through hospital stay, an average of 7 days
  death of a patient occurring during the index hospitalization of pulmonary embolism.

SECONDARY OUTCOMES:
procedural related complications | baseline, 72 hours post operation
  safety outcomes
major bleeding (as defined by BARC) | baseline, 72 hours post operation
  safety outcomes
hemoglobin change within 72 hours of the procedure | baseline, 72 hours post operation
  safety outcomes
change in the right ventricle to left ventricle ratio | baseline, 72 hours post operation
  procedural efficacy
mean pulmonary artery pressure | baseline, 72 hours post operation
  procedural efficacy
clinical deterioration and/or escalation to a bailout therapy | baseline, 72 hours post operation
  Clinical deterioration is defined by documented objective hemodynamic or respiratory worsening that is not present at the time of procedure, and will be reported as incidence.
  Bailout therapy is defined as use of an alternate treatment strategy not originally planned, and will be reported as incidence.
PE related mortality in 90 days | baseline, 90 days
  PE related mortality in 90 days

OTHER OUTCOMES:
90 days overall mortality rate | baseline, 90 days
  90 days mortality rate
PE recurrence by 90 days | baseline, 90 days
  recurrence of PE by 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided